CLINICAL TRIAL: NCT06129201
Title: Development of a Machine Learning Model for Nasopharyngeal Carcinoma Screening Based on Tongue Imaging: a Prospective Multicenter Cross-sectional Study
Brief Title: Development of a Machine Learning Model for Nasopharyngeal Carcinoma Screening Based on Tongue Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.ZYZLK.006
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Artificial Intelligence， Tongue Image
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training group: Experimental group: population of initially diagnosed nasopharyngeal carcinoma [600 people]; Control group: 2400 healthy individuals+nasopharyngeal disease patients+other tumors.
  Interventions: Other: Tongue image
- Validation group: Validation group: Experimental group: Nasopharyngeal cancer population [400 people]; Control group: 1600 healthy individuals+patients with nasopharyngeal diseases+other tumors.
  Interventions: Other: Tongue image

INTERVENTIONS:
Other: Tongue image — Using intelligent imaging devices to collect subject tongue images

SUMMARY:
Nasopharyngeal cancer is common in China, Southeast Asia, and North Africa, and is usually associated with Epstein-Barr virus (EBV) infection. Using EBV specific antibodies or EBV DNA screening can increase the proportion of patients diagnosed with early nasopharyngeal carcinoma from approximately 20% to over 70%. However, the application of nasopharyngeal carcinoma screening in clinical practice is hindered by low positive predictive values, even in areas where the EB virus is prevalent in China, the positive predictive value is only 4.8%. Therefore, there is an urgent need to identify new biomarkers or strategies with high sensitivity and positive predictive value for nasopharyngeal carcinoma screening.

A study published in the Lancet sub journal 《eClinicalMedicine》 in 2023 showed that a tongue image model based on machine learning can serve as a stable diagnostic method for gastric cancer (AUC=0.89), and has been clinically validated in multiple centers. This study inspires researchers to introduce artificial intelligence machine learning technology into the diagnosis and treatment of nasopharyngeal cancer.

In summary, this plan explores the establishment of tongue image machine learning models in nasopharyngeal carcinoma patients to help improve the positive predictive value of nasopharyngeal carcinoma screening.

DETAILED DESCRIPTION:
Nasopharyngeal cancer is common in China, Southeast Asia, and North Africa, and is generally associated with Epstein-Barr virus (EBV) infection. Using EBV specific antibodies or EBV DNA screening can increase the proportion of patients diagnosed with early nasopharyngeal carcinoma from approximately 20% to over 70%. In previous studies, researchers found that participants who underwent screening were more likely to achieve long-term survival after being diagnosed with nasopharyngeal carcinoma compared to the control group, and the risk of nasopharyngeal carcinoma specific death was lower among screened patients (relative risk 0.22). However, the application of nasopharyngeal carcinoma screening in clinical practice is hindered by low positive predictive values, even in areas where the EB virus is prevalent in China, the positive predictive value is only 4.8%. More than 95% of high-risk participants identified through primary serological screening underwent unnecessary and time-consuming clinical examinations and follow-up. The combination of various biomarkers, multi-step screening, and identification of new biomarkers are used to improve the performance of nasopharyngeal cancer screening strategies. However, the progress achieved so far is still unsatisfactory, characterized by low sensitivity, complex operation, or high cost. Therefore, there is an urgent need to identify new biomarkers or strategies with high sensitivity and positive predictive value for nasopharyngeal carcinoma screening.

In 《The New England Journal of Medicine》 in 2023, Professor Xia Ningshao's team reported on the identification and validation of anti BNLF2 total antibody (P85Ab) as a new serological biomarker for nasopharyngeal cancer screening.The sensitivity of P85-Ab nasopharyngeal carcinoma is 97.9%, with a positive predictive value of 10.0%. Furthermore, on the basis of P85-Ab positivity, if further detection of EB double antibodies (EBV nuclear antigen 1 [EBNA1]-IgA and EBV-specific viral capsid antigen [VCA]-IgA) is carried out, intermediate or medium high risk individuals with EB double antibodies can undergo nasopharyngoscopy examination, which can increase the positive predictive value of nasopharyngeal carcinoma screening to 29.6% -44.6%, that is, for every 2-3 nasopharyngoscopes performed, one case of nasopharyngeal carcinoma can be diagnosed. The sensitivity of this study is very high, but the positive predictive value is only 10%. Even when combined with traditional EB dual antibody monitoring and nasal endoscopy, one-third to one-half of non nasopharyngeal carcinoma patients still undergo unnecessary and time-consuming clinical examinations. Therefore, it is still necessary to explore simple and cost-effective methods to improve the strategy of positive predictive value for nasopharyngeal carcinoma screening.

A study published in the Lancet sub journal 《eClinicalMedicine》 in 2023 showed that a tongue image model based on machine learning can serve as a stable diagnostic method for gastric cancer (AUC=0.89), and has been clinically validated in multiple centers. This study inspires researchers to introduce artificial intelligence machine learning technology into the diagnosis and treatment of nasopharyngeal cancer.

In summary, this plan explores the establishment of tongue image machine learning models in nasopharyngeal carcinoma patients to help improve the positive predictive value of nasopharyngeal carcinoma screening.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients confirmed by histology/cytology
* Patients with nasopharyngeal carcinoma in the training group are initially diagnosed
* Subjects voluntarily participate in the study

Exclusion Criteria:

* Subjects taking medication or diet may affect their tongue image (such as aluminum magnesium carbonate, traditional Chinese medicine rhubarb, etc.)
* The researchers determined that the subjects had other factors that could force them to terminate the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study plans to include a training group consisting of 600 newly diagnosed nasopharyngeal carcinoma patients and 800 healthy individuals, as well as 800 individuals with common nasopharyngeal diseases and other tumors. According to the training group: validation group=6:4, configure the number of validation group members. There are approximately 5000 people in total.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of Diagnostic Model | 12 months
  Determine the screening effectiveness of the nasopharyngeal carcinoma tongue image model

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zeng, Doctor, Principal Investigator — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat sen University, Zhuhai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Background] Zeng Y, Zhang LG, Wu YC, Huang YS, Huang NQ, Li JY, Wang YB, Jiang MK, Fang Z, Meng NN. Prospective studies on nasopharyngeal carcinoma in Epstein-Barr virus IgA/VCA antibody-positive persons in Wuzhou City, China. Int J Cancer. 1985 Nov 15;36(5):545-7. doi: 10.1002/ijc.2910360505. PMID 4055129
- [Background] Liu Z, Ji MF, Huang QH, Fang F, Liu Q, Jia WH, Guo X, Xie SH, Chen F, Liu Y, Mo HY, Liu WL, Yu YL, Cheng WM, Yang YY, Wu BH, Wei KR, Ling W, Lin X, Lin EH, Ye W, Hong MH, Zeng YX, Cao SM. Two Epstein-Barr virus-related serologic antibody tests in nasopharyngeal carcinoma screening: results from the initial phase of a cluster randomized controlled trial in Southern China. Am J Epidemiol. 2013 Feb 1;177(3):242-50. doi: 10.1093/aje/kws404. Epub 2012 Dec 19. PMID 23255783
- [Background] Ji MF, Sheng W, Cheng WM, Ng MH, Wu BH, Yu X, Wei KR, Li FG, Lian SF, Wang PP, Quan W, Deng L, Li XH, Liu XD, Xie YL, Huang SJ, Ge SX, Huang SL, Liang XJ, He SM, Huang HW, Xia SL, Ng PS, Chen HL, Xie SH, Liu Q, Hong MH, Ma J, Yuan Y, Xia NS, Zhang J, Cao SM. Incidence and mortality of nasopharyngeal carcinoma: interim analysis of a cluster randomized controlled screening trial (PRO-NPC-001) in southern China. Ann Oncol. 2019 Oct 1;30(10):1630-1637. doi: 10.1093/annonc/mdz231. PMID 31373615
- [Background] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880
- [Background] Miller JA, Le QT, Pinsky BA, Wang H. Cost-Effectiveness of Nasopharyngeal Carcinoma Screening With Epstein-Barr Virus Polymerase Chain Reaction or Serology in High-Incidence Populations Worldwide. J Natl Cancer Inst. 2021 Jul 1;113(7):852-862. doi: 10.1093/jnci/djaa198. PMID 33351145
- [Background] Simon J, Liu Z, Brenner N, Yu KJ, Hsu WL, Wang CP, Chien YC, Coghill AE, Chen CJ, Butt J, Proietti C, Doolan DL, Hildesheim A, Waterboer T. Validation of an Epstein-Barr Virus Antibody Risk Stratification Signature for Nasopharyngeal Carcinoma by Use of Multiplex Serology. J Clin Microbiol. 2020 Apr 23;58(5):e00077-20. doi: 10.1128/JCM.00077-20. Print 2020 Apr 23. PMID 32102852
- [Background] Coghill AE, Pfeiffer RM, Proietti C, Hsu WL, Chien YC, Lekieffre L, Krause L, Teng A, Pablo J, Yu KJ, Lou PJ, Wang CP, Liu Z, Chen CJ, Middeldorp J, Mulvenna J, Bethony J, Hildesheim A, Doolan DL. Identification of a Novel, EBV-Based Antibody Risk Stratification Signature for Early Detection of Nasopharyngeal Carcinoma in Taiwan. Clin Cancer Res. 2018 Mar 15;24(6):1305-1314. doi: 10.1158/1078-0432.CCR-17-1929. Epub 2018 Jan 4. PMID 29301829
- [Background] He YQ, Wang TM, Ji M, Mai ZM, Tang M, Wang R, Zhou Y, Zheng Y, Xiao R, Yang D, Wu Z, Deng C, Zhang J, Xue W, Dong S, Zhan J, Cai Y, Li F, Wu B, Liao Y, Zhou T, Zheng M, Jia Y, Li D, Cao L, Yuan L, Zhang W, Luo L, Tong X, Wu Y, Li X, Zhang P, Zheng X, Zhang S, Hu Y, Qin W, Deng B, Liang X, Fan P, Feng Y, Song J, Xie SH, Chang ET, Zhang Z, Huang G, Xu M, Feng L, Jin G, Bei J, Cao S, Liu Q, Kozlakidis Z, Mai H, Sun Y, Ma J, Hu Z, Liu J, Lung ML, Adami HO, Shen H, Ye W, Lam TH, Zeng YX, Jia WH. A polygenic risk score for nasopharyngeal carcinoma shows potential for risk stratification and personalized screening. Nat Commun. 2022 Apr 12;13(1):1966. doi: 10.1038/s41467-022-29570-4. PMID 35414057
- [Background] Zhou X, Cao SM, Cai YL, Zhang X, Zhang S, Feng GF, Chen Y, Feng QS, Chen Y, Chang ET, Liu Z, Adami HO, Liu J, Ye W, Zhang Z, Zeng YX, Xu M. A comprehensive risk score for effective risk stratification and screening of nasopharyngeal carcinoma. Nat Commun. 2021 Aug 31;12(1):5189. doi: 10.1038/s41467-021-25402-z. PMID 34465768
- [Background] Lam WKJ, Jiang P, Chan KCA, Cheng SH, Zhang H, Peng W, Tse OYO, Tong YK, Gai W, Zee BCY, Ma BBY, Hui EP, Chan ATC, Woo JKS, Chiu RWK, Lo YMD. Sequencing-based counting and size profiling of plasma Epstein-Barr virus DNA enhance population screening of nasopharyngeal carcinoma. Proc Natl Acad Sci U S A. 2018 May 29;115(22):E5115-E5124. doi: 10.1073/pnas.1804184115. Epub 2018 May 14. PMID 29760067
- [Background] Lam WKJ, Jiang P, Chan KCA, Peng W, Shang H, Heung MMS, Cheng SH, Zhang H, Tse OYO, Raghupathy R, Ma BBY, Hui EP, Chan ATC, Woo JKS, Chiu RWK, Lo YMD. Methylation analysis of plasma DNA informs etiologies of Epstein-Barr virus-associated diseases. Nat Commun. 2019 Jul 22;10(1):3256. doi: 10.1038/s41467-019-11226-5. PMID 31332191
- [Background] Chen GH, Liu Z, Yu KJ, Coghill AE, Chen XX, Xie SH, Lin DF, Huang QH, Lu YQ, Ling W, Lin CY, Lu ZJ, Fan YY, Tang LQ, Sampson JN, Li H, King AD, Middeldorp JM, Hildesheim A, Cao SM. Utility of Epstein-Barr Virus DNA in Nasopharynx Swabs as a Reflex Test to Triage Seropositive Individuals in Nasopharyngeal Carcinoma Screening Programs. Clin Chem. 2022 Jul 3;68(7):953-962. doi: 10.1093/clinchem/hvac032. PMID 35325087
- [Background] Li T, Li F, Guo X, Hong C, Yu X, Wu B, Lian S, Song L, Tang J, Wen S, Gao K, Hao M, Cheng W, Su Y, Zhang S, Huang S, Fang M, Wang Y, Ng MH, Chen H, Luo W, Ge S, Zhang J, Xia N, Ji M. Anti-Epstein-Barr Virus BNLF2b for Mass Screening for Nasopharyngeal Cancer. N Engl J Med. 2023 Aug 31;389(9):808-819. doi: 10.1056/NEJMoa2301496. PMID 37646678
- [Background] Yuan L, Yang L, Zhang S, Xu Z, Qin J, Shi Y, Yu P, Wang Y, Bao Z, Xia Y, Sun J, He W, Chen T, Chen X, Hu C, Zhang Y, Dong C, Zhao P, Wang Y, Jiang N, Lv B, Xue Y, Jiao B, Gao H, Chai K, Li J, Wang H, Wang X, Guan X, Liu X, Zhao G, Zheng Z, Yan J, Yu H, Chen L, Ye Z, You H, Bao Y, Cheng X, Zhao P, Wang L, Zeng W, Tian Y, Chen M, You Y, Yuan G, Ruan H, Gao X, Xu J, Xu H, Du L, Zhang S, Fu H, Cheng X. Development of a tongue image-based machine learning tool for the diagnosis of gastric cancer: a prospective multicentre clinical cohort study. EClinicalMedicine. 2023 Feb 6;57:101834. doi: 10.1016/j.eclinm.2023.101834. eCollection 2023 Mar. PMID 36825238